CLINICAL TRIAL: NCT05139303
Title: Efficacy of the OrthoApnea NOA® Mandibular Advancement Device in the Management of Obstructive Sleep Apnea. Clinical Trial and Retrospective Comparison Study.
Brief Title: Efficacy of the OrthoApnea NOA® Mandibular Advancement Device in the Management of Obstructive Sleep Apnea.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isabel Moreno Hay (Other)
Responsible Party: Sponsor-Investigator, Isabel Moreno Hay, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 71295
Record Dates: First submitted 2021-11-04; First posted 2021-12-01 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA; Obstructive sleep apnea; mandibular advancement device; oral appliance
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MAD therapy (Experimental): An NOA® appliance (Orthoapnea S.L., Malaga, Spain) was custom made for each participant at 50% from maximum protrusion.
  Interventions: Device: Orthoapnea NOA®

INTERVENTIONS:
Device: Orthoapnea NOA® — The efficacy of the appliance for the management of OSA will be stablished based on two criteria. Criterion I: > 50% reduction of AHI/RDI. Criterion II: AHI/RDI < 5 events/hour or <15 events/hour with a significative reduction of OSA associates symptoms as defined before. Therapeutic failure will be established when at 100% of advancement of the device, there is less than 50% of reduction of the AHI/RDI with a residual AHI/RDI >5 events/hour with OSA associates symptoms.

SUMMARY:
The objective of this study is to assess the efficacy of the Orthoapnea NOA® mandibular advancement device and describe the percentage of advancement (%) needed to reach efficacy, and to retrospectively compare with other MAD designs in the management of obstructive sleep apnea. Additionally, to describe patient compliance and adherence to the therapy with the Orthoapnea NOA® device, and to assess the incidence and prevalence of signs, symptoms, and diagnosis of temporomandibular disorders (TMD) associated to the use of the Orthoapnea NOA® mandibular advancement device.

DETAILED DESCRIPTION:
Participants were recruited consecutively from patients referred by a board certified sleep physician to the Orofacial Pain Clinic (University of Kentucky, Lexington, Kentucky, USA) for the management of OSA with a mandibular advancement device. An NOA® appliance (Orthoapnea S.L., Malaga, Spain) was custom made for each participant. Digital impressions (scanner 3Shape TRIOS® 3, Copenhagen, Denmark), protrusive records at 50% from maximum protrusion (using a 5 mm fork and George GaugeTM, Great Lakes Dental Technologies, Tonawanda, NY, USA), and clinical pictures were obtained following the protocol recommended by the manufacturer. Maximum mouth opening was measured by adding the interincisal distance to the overbite (in millimeters, using TheraBite® Range of Motion ruler, Great Lakes Dental Technologies, Tonawanda, NY, USA). The MAD was fabricated at an initial protrusion of 50%, with subsequent progressive mandibular components of additional 10% of protrusion up to 100% of the maximum protrusive range. Lastly, a full coverage morning deprogrammer (TAP® AM Aligner, World Class Technology Corp., McMinniville, OR, USA) was fabricated for all the participants to be used for 10 minutes upon removal of the MAD. Follow up visits were scheduled every two weeks and measures of compliance, sleep parameters, pain, headaches, TMD and side effects were monitored.

ELIGIBILITY:
Inclusion Criteria:

* Age: >18 and <80 years old.
* No history of previous use of a MAD.
* Diagnosis of OSA by a sleep physician based on a PSG or HSAT (done >12 months before evaluation date or > 12 months with >10% variation of BMI).
* Upon clinical examination: >8 teeth per arch; range of anteroposterior mandibular mobility >5 mm.
* Informed consent to participate in the study.

Exclusion Criteria:

* Patients with concomitant diagnosed sleep disorders (i.e. insomnia, narcolepsy, restless legs syndrome, rapid eye movement sleep behavior disorder).
* History of previous allergic reaction to the appliance material (Polyamide 12).
* Patients using combination therapy for the management of OSA (i.e. PAP therapy or positional therapy).
* Upon clinical examination: periodontal disease (>4 mm on periodontal probing, with bleeding on probing, visual signs of periodontal inflammation); tooth horizontal mobility >1 mm, vertical mobility, and unfavorable crown to root ratio; open cavities, loose or fractured restorations, or patient undergoing restorative dental treatments.
* Exaggerated gag reflex.
* Lack of coordination or dexterity.
* Inadequate English comprehension.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Moreno Hay, Principal Investigator — University of Kentucky
Locations (1):
- Orofacial Pain Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited consecutively from patients referred to the Orofacial Pain Clinic for the management of obstructive sleep apnea.
Pre-assignment Details: 4 participants were excluded, three of them did not report back to their follow up appointment and one could not tolerate the intervention.
Groups:
- Retrospective MAD: Archival data were extracted from a database of patients that started MAD therapy for OSA between January of 2010 and August of 2021 at the same clinic and that had a second sleep study performed to assess the effectiveness of the MAD.
Period: Overall Study
Arm/Group | MAD Therapy | Retrospective MAD
Started | 37 | 59
Completed | 33 | 59
Not Completed | 4 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MAD Therapy | Retrospective MAD | Total
Number analyzed (Participants) | 33 | 59 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.36 (15.76) | 59.03 (10.31) | 55.70 (13.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 27 | 48
  Male | 12 | 32 | 44
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI) is calculated by using weight in kilograms (kg) divided by the square of height in meters (m2).
  kg/m^2 | 30.57 (5.72) | 31.93 (7.07) | 31.25 (6.40)
Apnea Hypopnea Index (AHI) [Mean (Standard Deviation); unit: events/hour] — Apnea Hypopnea Index (AHI) is calculated by adding the total amount of apneas and hypopneas during the study and dividing that number by total sleep time.
  events/hour | 15.34 (11.27) | 23.46 (16.76) | 19.40 (14.02)
Minimum oxygen saturation [Mean (Standard Deviation); unit: % of oxygen saturation] — A pulse oximeter is used to calculate the minimum oxygen saturation by measuring light wavelengths to determine the ratio of the current levels of oxygenated hemoglobin to deoxygenated hemoglobin.
  % of oxygen saturation | 84.91 (4.36) | 82.28 (6.42) | 83.60 (5.39)

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Number of Participants That Responded to the Mandibular Advancement Device (MAD)
Description: Assessment of efficacy of the device: After delivery, the MAD will be advanced 10% every 2 weeks until maximum therapeutic benefit. Sleep parameters (apnea hypopnea index (AHI) and minimum oxygen saturation) will be extracted from the initial polysomnography (PSG), and from a final confirmatory home sleep apnea test. The efficacy will be stablished based on: Criterion I: > 50% reduction of AHI; Criterion II: AHI < 5 events/hour or <15 events/hour with a significant reduction of obstructive sleep apnea (OSA) associated symptoms.
Time Frame: 16 weeks.
Measure: Number; unit: participants
Arm/Group | MAD Therapy | Retrospective MAD
Number analyzed (Participants) | 33 | 59
participants
  Criterion 1 | 26 | 37
  Criterion 2 | 30 | 20
Statistical Analysis 1: Comparison: MAD Therapy; Test type: Other; p < 0.05, Chi-squared

2. Primary Outcome: % of Advancement of the Jaw Needed to Achieve Efficacy With the Use of the Mandibular Advancement Device (MAD) Based on the Success Criterion I and II
Description: Criterion I: > 50% reduction of AHI/RDI. Criterion II: AHI/RDI < 5 events/hour or <15 events/hour with a significative reduction of OSA associates symptoms as defined before. Therapeutic failure will be established when at 100% of advancement of the device, there is less than 50% of reduction of the AHI/RDI with a residual AHI/RDI >5 events/hour with OSA associates symptoms.
Time Frame: 16 weeks
Population: Number of participants analyzed were those succeeding for Criterion 1 and Criterion 2
Measure: Mean (Standard Deviation); unit: percentage of mandibular protrusion
Groups:
- MAD Therapy: The efficacy of the appliance for the management of OSA will be stablished based on two criteria. Criterion I: > 50% reduction of AHI/RDI. Criterion II: AHI/RDI < 5 events/hour or <15 events/hour with a significative reduction of OSA associates symptoms as defined before. Therapeutic failure will be established when at 100% of advancement of the device, there is less than 50% of reduction of the AHI/RDI with a residual AHI/RDI >5 events/hour with OSA associates symptoms.
Arm/Group | MAD Therapy | Retrospective MAD
Number analyzed (Participants) | 33 | 59
percentage of mandibular protrusion
  Criterion I: number analyzed (Participants) | 26 | 37
  Criterion I | 80 (10.2) | 88.73 (14)
  Criterion II: number analyzed (Participants) | 30 | 20
  Criterion II | 75.33 (10.08) | 89.59 (15.91)

3. Secondary Outcome: Number of Participants Compliant to the Mandibular Advancement Device (MAD)
Description: The self-reported use of mandibular advancement device (MAD) was assessed at each follow-up via questionnaire on a five-point checklist (number hours per night and nights per week). Compliance was defined as wearing the appliance for ≥4 hours per night during at least 70% of the nights.
Time Frame: 16 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | MAD Therapy | Retrospective MAD
Number analyzed (Participants) | 33 | 59
Participants | 33 | 59

4. Other Pre Specified Outcome: Incidence of Temporomandibular Disorders (TMD) Associated to the Use of the Mandibular Advancement Device (MAD). the Use of the Orthoapnea NOA® Mandibular Advancement Device.
Description: Number of participants that develop of signs, symptoms of TMD will be assessed following the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD).
Time Frame: 16 weeks.
Population: Data were not collected from the retrospective study group for this measure
Measure: Count of Participants; unit: Participants
Arm/Group | MAD Therapy | Retrospective MAD
Number analyzed (Participants) | 33 | 0
Participants | 18 |

ADVERSE EVENTS:
Time Frame: From enrollment to the end of treatment at week 16. Participants were assessed every visit (every 2 weeks) from delivery of the mandibular advancement device until the end of follow up (week 16).
Description: The use of mandibular advancement devices for the management of obstructive sleep apnea are non invasive and reversible; adverse event data were not collected from the retrospective MAD group
Arm/Group | MAD Therapy
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 1/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MAD Therapy (N=33)
Jaw pain upon use of the mandibular advancement device (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT05139303/Prot_SAP_000.pdf